CLINICAL TRIAL: NCT07329699
Title: Artificial Intelligence-Driven Angiography-Based Fractional Flow Reserve Versus Invasive Fractional Flow Reserve-Guided PCI
Brief Title: Artificial Intelligence-Driven Medipixel Fractional Flow Reserve Versus Invasive Fractional Flow Reserve-Guided PCI Trial (AIM-FFR Trial)
Acronym: AIM-FFR
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Samsung Medical Center (Other)
Collaborators: Chonnam National University Hospital (Other); Seoul National University Bundang Hospital (Other); Chung-Ang University Gwangmyeong Hospital (Other); The Catholic University of Korea (Other); Keimyung University Dongsan Medical Center (Other); Wonju Severance Christian Hospital (Other); SMG-SNU Boramae Medical Center (Other); Kangbuk Samsung Hospital, Sungkyunkwan University (Other); Korea University Guro Hospital (Other); Inje University Ilsan Paik Hospital (Other); International St. Mary's Hospital (Unknown); Kyungpook National University Hospital (Other); Korea University Anam Hospital (Other); Ajou University School of Medicine (Other); Changwon Patima Hospital (Unknown); Bundang CHA Hospital (Other); Ulsan University Hospital (Other); Gachon University Gil Medical Center (Other); Inje University Haeundae Paik Hospital (Other); Gyeongsang National University Changwon Hospital (Other); Wonkwang University Hospital (Other)
Responsible Party: Principal Investigator, Joo Myung Lee, Associate Professor, Samsung Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SMC19810222
Record Dates: First submitted 2025-12-23; First posted 2026-01-09 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Coronary Artery Disease; Chronic Coronary Syndrome; Acute Coronary Syndrome
Keywords: Coronary artery stenosis; Fractional flow reserve; Prognosis
MeSH Terms: conditions — Coronary Artery Disease; Acute Coronary Syndrome; Coronary Stenosis

STUDY DESIGN:
Intervention Model Description: A prospective, multi-center, open-label, randomized controlled, non-inferiority trial.
Who Masked: Participant, Outcomes Assessor
Masking Description: Patients will be blinded to the assigned groups. Clinical events will be independently adjudicated by independent Clinical Events Adjudication Committee.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MPFFR-guided PCI group (Experimental): In patients randomized to artificial intelligence-driven angiography-based fractional flow reserve (MPFFR)-guided PCI group, MPFFR analysis will be performed using MPFFR-1000 version 2.1.0 (Medipixel Inc., Seoul, Korea). Manual correction can be applied when necessary, however, it will be strongly discouraged by the study protocols. Treatment decisions will be made based on site-measured MPFFR value.
  Functionally significant stenosis will be defined as MPFFR≤0.80. For lesions with MPFFR≤0.80, PCI will be recommended under current guidelines, however, final decision regarding PCI will be at the discretion of operators. In the MPFFR-guided PCI group, on-site MPFFR value will be used in decision making of revascularization. If PCI is not performed for lesions with MPFFR≤0.80, the specific reasons will be collected in electronic case report form. For lesions with MPFFR>0.80, PCI will be deferred.
  Interventions: Diagnostic Test: MPFFR or Invasive FFR
- Invasive FFR-guided PCI group (Active Comparator): All invasive FFR measurements will be performed after diagnostic coronary angiography according to a standardized protocol as previously described. A pressure-temperature sensor guide wire (Abbott Vascular, Santa Clara, CA, USA) is positioned at the distal segment of the target lesion. To induce maximal hyperemia state, intravenous infusion of adenosine (140μg/kg/min through a peripheral vein) or intracoronary injection of nicorandil (2mg) will be used. In the presence of drift greater than 0.03 FFR unit, pressure wire will be re-equalized and FFR will be measured again.
  Functionally significant stenosis will be defined as FFR≤0.80. For lesions with FFR≤0.80, PCI will be recommended under current guidelines, however, final decision regarding PCI will be at the discretion of operators. If PCI is not performed for lesions with FFR≤0.80, the specific reasons will be collected in electronic case report form. For lesions with FFR>0.80, PCI will be deferred.
  Interventions: Diagnostic Test: MPFFR or Invasive FFR

INTERVENTIONS:
Diagnostic Test: MPFFR or Invasive FFR — Functionally significant stenosis will be defined as MPFFR≤0.80 or FFR≤0.80. For lesions with MPFFR≤0.80 or FFR≤0.80, PCI will be recommended under current guidelines, however, final decision regarding PCI will be at the discretion of operators. In the MPFFR-guided PCI group, on-site MPFFR value will be used in decision making of revascularization. If PCI is not performed for lesions with MPFFR≤0.80 or FFR≤0.80, the specific reasons will be collected in electronic case report form. For lesions with MPFFR>0.80 or FFR>0.80, PCI will be deferred.

SUMMARY:
The AIM-FFR trial is a prospective, multi-center, open-label, randomized controlled, non-inferiority trial. The current trial will evaluate non-inferiority of MPFFR-guided PCI, compared with invasive FFR-guided PCI in patients with coronary artery disease.

DETAILED DESCRIPTION:
Fractional Flow Reserve (FFR) has been established as the gold standard for determining the functional significance of coronary artery stenosis. Current guidelines have classified FFR as a Class IA recommendation for the assessment of intermediate coronary artery lesions. However, FFR remains underused in daily clinical practice, due to requirement for pressure wire use, hyperemia induction, or prolonged procedural time.

To overcome these limitations, angiography-derived computation of FFR have been widely adopted as wire-free alternatives. These technologies enable functional assessment of coronary stenosis without pressure wires, providing a less invasive and more comfortable alternative to wire-based FFR. Multiple modalities have shown reasonable diagnostic accuracy to predict FFR≤0.80. Among them, Quantitative Flow Ratio (QFR)-guided percutaneous coronary intervention (PCI) demonstrated superior clinical outcome than angiography-guided PCI. Based on these results, QFR-guided PCI is supported by class 1B recommendation from European Society of Cardiology guideline. Nevertheless, angiography-derived FFR also has limitations, primarily related to the technical and workflow demands of the process. Computation of angiography-derived FFR typically requires vessel segmentation, correspondence marking, and 3-dimensional reconstruction from angiographic images, which are time-consuming and subject to operator-dependent variability.

Indeed, recent data shows limitations of angiography-based FFR computation. Study by Ninomiya et al. evaluated five different angiography-derived FFR methods (QFR, vFFR from Pie Medical Imaging, caFFR from Rainmed Ltd, 2D-µFR, and 3D-µFR from Pulse Medical Imaging Technology). Although these angiography-derived FFR methods provided higher discrimination than angiographic stenosis severity to discriminate functionally significant stenosis defined by FFR≤0.80 or instantaneous wave-free ratio≤0.89, the AUC ranged from 0.65 to 0.75. Furthermore, recent FAVOR III Europe trial showed that QFR-guided strategy did not meet non-inferiority to FFR-guided strategy in terms of a composite of death, myocardial infarction, and unplanned revascularization at 12 months. These results support invasive FFR-guided strategy is gold standard method.

Recent advances in Artificial Intelligence (AI) have led to development of automated tools for cardiovascular diagnostics, improving both accuracy and workflow efficiency. The AI-driven angiography-based FFR (Medipixel FFR [MPFFR]) has been developed utilizing AI-based fully automated quantitative coronary angiography (AI-QCA). MPFFR utilizes automated frame selection, AI-based contouring, and real-time modeling, allowing for rapid and accurate physiological assessment without manual segmentation. In previous validation study conducted in Korea (599 vessels from 452 patients who underwent clinically indicated FFR measurement from 5 university hospitals in Korea), Mean analysis time of MPFFR was 12.5±1.7 seconds and manual correction was needed in 32 vessels (5.3%). MPFFR showed similar diagnostic performance with QFR (correlation with FFR; MPFFR vs. QFR: R=0.885 vs. R=0.860, P for comparison=0.011; area under curve to predict FFR≤0.80; 0.949 vs. 0.953, P for comparison=0.631). At a median follow-up of 2 years (interquartile range, 1.6 to 2.6 years), patients with MPFFR≤0.80 had higher risk of target vessel failure than those with MPFFR>0.80 (4.5% vs. 0.8%; adjusted HR, 5.94; 95% CI, 1.27-27.91; P=0.024). C-index to predict target vessel failure was comparable between MPFFR and QFR (0.770 vs. 0.753, P for comparison=0.469).

However, whether MPFFR-guided PCI can be used in daily practice still needs to be validated by randomized controlled trial using invasive FFR-guided PCI as reference standard. On this background, the current trial aims to compare clinical outcomes between MPFFR-guided PCI and invasive FFR-guided PCI in patients with coronary artery disease.

ELIGIBILITY:
Inclusion Criteria:

1. Subject must be at least 19 years of age
2. Eligible for coronary angiography and/or percutaneous coronary intervention.
3. Chronic coronary syndrome or acute coronary syndrome (non-culprit vessels only)
4. Coronary artery disease in one or more native major epicardial vessels or their branches with reference vessel diameter of at least 2.5mm and with visually assessed coronary stenosis in which the physiological severity of the lesion is questionable (typically 40-90% diameter stenosis).
5. Subject who is able to understand risks, benefits and treatment alternatives and sign informed consent voluntarily.

Exclusion Criteria:

1. Patients unable to provide informed consent
2. Patients with known intolerance to aspirin, P2Y12 inhibitors, or components of drug-eluting stents and drug-coated balloons
3. Patients with coronary artery bypass grafting
4. Patients who have non-cardiac co-morbid conditions with life expectancy <1 year
5. Patients with cardiogenic shock or cardiac arrest
6. Patients with severe left ventricular systolic dysfunction (ejection fraction <30%)
7. Patients with severe valvular heart disease requiring open heart surgery
8. Pregnant or lactating women
9. Angiographic exclusion criteria

   * Culprit vessel of patients with ST-elevation myocardial infarction (target lesions in non-culprit vessel can be enrolled)
   * Chronic total occlusion (target lesions in vessels without chronic total occlusion can be enrolled)
   * Ostial stenosis in left man coronary artery or right coronary artery
   * Severe tortuosity of any target vessel
   * Severe overlap in the stenosed segment
   * Poor image quality precluding identification of vessel contours

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2100 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2028-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Major adverse cardiac events (MACE) | 1 year after last patient enrollment
  a composite of death from any causes, non-fatal myocardial infarction [MI], and clinically indicated unplanned revascularization

SECONDARY OUTCOMES:
All-cause death | 1 year after last patient enrollment
  All-cause death (defined by Academic Research Consortium [ARC] II definition)
Cardiovascular death | 1 year after last patient enrollment
  Cardiovascular death (defined by Academic Research Consortium [ARC] II definition)
Non-fatal myocardial infarction (MI) | 1 year after last patient enrollment
  Non-fatal MI (according to the Fourth universal definition of MI)
Target vessel-related MI | 1 year after last patient enrollment
  Target vessel-related MI (Target vessel denotes vessels with initially interrogated by MPFFR or invasive FFR)
Non-target vessel-related MI | 1 year after last patient enrollment
  Non-target vessel-related MI (Target vessel denotes vessels with initially interrogated by MPFFR or invasive FFR)
Clinically indicated unplanned revascularization | 1 year after last patient enrollment
  Clinically indicated unplanned revascularization (defined by Academic Research Consortium [ARC] II definition)
Clinically indicated target vessel revascularization | 1 year after last patient enrollment
  Clinically indicated target vessel revascularization (Target vessel denotes vessels with initially interrogated by MPFFR or invasive FFR)
Clinically indicated non-target vessel repeat revascularization | 1 year after last patient enrollment
  Clinically indicated non-target vessel repeat revascularization (Target vessel denotes vessels with initially interrogated by MPFFR or invasive FFR)
Vessel or Stent thrombosis | 1 year after last patient enrollment
  Vessel or Stent thrombosis (definite thrombosis defined by Academic Research Consortium [ARC] II definition)
Cardiovascular death or target vessel-related MI | 1 year after last patient enrollment
  A composite of Cardiovascular death or target vessel-related MI
Target vessel failure | 1 year after last patient enrollment
  Target vessel failure (TVF, a composite of cardiovascular death, target vessel-related MI, and clinically indicated target vessel revascularization)
Bleeding according to BARC definition | 1 year after last patient enrollment
  Bleeding according to BARC definition
Cerebrovascular accident (CVA) | 1 year after last patient enrollment
  Cerebrovascular accident (CVA) including ischemic stroke, hemorrhagic stroke, or transient ischemic attack (TIA)
Contrast volume (including both diagnostic angiography and PCI) | immediately after the intervention/procedure
  Contrast volume (including both diagnostic angiography and PCI)
Procedure time of MPFFR or invasive FFR measurement | immediately after the intervention/procedure
  Procedure time of MPFFR or invasive FFR measurement
Procedure time including the decision-making time for PCI following coronary angiography | immediately after the intervention/procedure
  Procedure time including the decision-making time for PCI following coronary angiography
Number of lesions interrogated | immediately after the intervention/procedure
  Number of lesions interrogated by MPFFR or invasive FFR
Number of used stents or drug-coated balloons | immediately after the intervention/procedure
  Number of used stents or drug-coated balloons

CONTACTS AND LOCATIONS:
Overall Officials: Joo Myung Lee, MD, MPH, PhD, Principal Investigator — Samsung Medical Center
Locations (25):
- South Korea (25):
  - Korea University Anam Hospital, Seoul, Select State
  - Inje University Haeundae Paik Hospital, Busan
  - Changwon Fatima Hospital, Changwon
  - Gyeongsang National University Changwon Hospital, Changwon
  - Keimyung University Dongsan Hospital, Daegu
  - Kyungpook National University Hospital, Daegu
  - Chonnam National University Hospital, Chonnam National University Medical School, Gwangju
  - Chung-Ang University Gwangmyeong Hospital, Gwangmyeong
  - CHA Bundang Medical Center, Gyeonggi-do
  - Wonkwang University Hospital, Iksan
  - Inje University College of Medicine, Ilsan Paik Hospital, Ilsan
  - Gachon University Gil Medical Center, Incheon
  - Inha University Hospital, Incheon
  - International St. Mary's Hospital, Incheon
  - Presbyterian Medical Center, Jeonju
  - Gyeongsang National University Hospital, Jinju
  - Seoul National University Bundang Hospital, Seongnam
  - Samsung Medical Center, Seoul
  - Kangbuk Samsung Hospital, Sungkyunkwan University School of Medicine, Seoul
  - Korea University Guro Hospital, Seoul
  - Seoul National University Boramae Medical Center, Seoul
  - Ajou University Hospital, Suwon
  - Uijeongbu ST. Mary's Hospital, Uijeongbu-si
  - Ulsan University Hospital, Ulsan
  - Wonju Severance Christian Hospital, Wŏnju

IPD SHARING:
Plan to Share IPD: Yes
Reseanable request will be reviwed by the Executive Committee.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: After publication of primary report and prespecified subgroup analysis.
Access Criteria: Reseanable request will be reviwed by the Executive Committee.